CLINICAL TRIAL: NCT00040534
Title: Safety and Tolerability Study of Farnesyl Protein Transferase Inhibitor in Combination With Gemcitabine and Cisplatin in Advanced Cancer (Study P01499)(TERMINATED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01499
Record Dates: First submitted 2002-06-28; First posted 2002-07-01 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms
Keywords: Advanced Cancer
MeSH Terms: conditions — Neoplasms | interventions — 2-(2-oxo-2-((3,7,11-trimethyl-2,6,10-dodecatrienyl)oxy)aminoethyl)phosphonic acid, (2,2-dimethyl-1-oxopropoxy)methyl ester sodium

INTERVENTIONS:
Drug: Farnesyl Protein Transferase Inhibitor

SUMMARY:
The purpose of this study is to determine the safety and tolerability of an oral Farnesyl Protein Transferase

Inhibitor (SCH 66336) when given in combination with Gemcitabine and Cisplatin in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer for which there is no treatment available which would have a reasonable chance of disease palliation or cure
* Age greater than or equal to 18.
* SWOG performance Status less than or equal to 2.
* Meets protocol requirements for specified laboratory values.
* Written informed consent and cooperation of patient.

Exclusion Criteria:

* Prior treatment with an FPTI
* Knowledge of intracranial metastases or carcinomatous meningitis.
* Poor medical risks because of nonmalignant systemic disease or uncontrolled active infection.
* Medical conditions that would interfere with taking oral medications.
* Significant uncontrolled diarrhea.
* Chemotherapy, radiotherapy or major surgery within 4 weeks; full recovery from prior treatment.
* Concomitant use of CYP3A inhibitors/inducers per protocol.
* Known HIV positivity or AIDS-related illness.
* Pregnant or nursing women.
* Men or women of childbearing potential who are not using an effective method of contraception.
* Concurrent chemotherapy, hormonal therapy, radiotherapy or immunotherapy.
* QTc prolongation (>440 msecs) at baseline.
* Patients with previous high-dose therapy requiring stem cell rescue or bone marrow transplant, or irradiation to >30% of bone marrow-containing areas.
* Patients that have received Mitomycin-C or nitrosoureas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

REFERENCES:
- [Result] Chow LQ, Eckhardt SG, O'Bryant CL, Schultz MK, Morrow M, Grolnic S, Basche M, Gore L. A phase I safety, pharmacological, and biological study of the farnesyl protein transferase inhibitor, lonafarnib (SCH 663366), in combination with cisplatin and gemcitabine in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2008 Sep;62(4):631-46. doi: 10.1007/s00280-007-0646-x. Epub 2007 Dec 6. PMID 18058098